CLINICAL TRIAL: NCT04475523
Title: Phase 1 Study of CI-8993 Anti-VISTA Antibody in Patients With Advanced Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Curis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI-8993-101
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Solid Tumor

STUDY DESIGN:
Intervention Model Description: Each patient will be administered a step-dose of CI-8993. If a patient experiences a DLT following the step dose, treatment will be discontinued for that patient. If there are no safety concerns following the step dose, the patient will receive the first full dose of CI-8993 a week later. If none of the 3 patients in each cohort (or 1 in 6 patients) experiences a DLT during the first cycle (28 days following the first full dose), the SRC may clear the next dose level for enrollment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CI-8993 dose escalation (Experimental): Patients will be administered CI-8993 intravenously at a planned infusion rate over 2 hours at planned step-doses and subsequent full doses. The planned schedule of administration is every 2 weeks. The MTD of full doses of CI-8993 will be determined based on the occurrence of DLTs 28 days from the first full dose. Eligible patients may receive CI-8993 at the dose and schedule, according to their assigned cohorts, until disease progression or unacceptable toxicity.
  Interventions: Drug: CI-8993

INTERVENTIONS:
Drug: CI-8993 — CI-8993 is a fully human immunoglobulin (Ig) G1κ monoclonal antibody (mAb) against the VISTA ligand

SUMMARY:
This is a phase 1, open-label, multicenter dose-escalation study to determine the RP2D of CI 8993 for administration to patients with relapsed/refractory solid tumors by evaluating the safety and tolerability and characterizing the PK, PD, and anti cancer activity of CI-8993 in this population.

DETAILED DESCRIPTION:
The plan is to enroll approximately 50 patients with metastatic or unresectable solid tumor malignancy (non-lymphoma) that is considered relapsed and/or refractory to prior therapy into specific dose cohorts to determine the maximum tolerated dose (MTD) of full doses of CI-8993, based on the occurrence of dose limiting toxicities (DLTs) 28 days from the first full dose. Administration is every 2 weeks. To assure patient safety, each patient will receive an initial low dose of CI-8993 (step-dose) one week prior to their first full dose.

A Safety Review Committee (SRC) will review all safety data and make cohort escalation/de-escalation decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be ≥18 years of age
2. Patients must have the following disease related criteria:

   * any type of solid tumor malignancy (non-lymphoma) that is metastatic or unresectable and considered relapsed and/or refractory to prior therapy
   * must have evaluable disease.
   * Archival formalin-fixed, paraffin-embedded (FFPE) tumor tissue
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Adequate organ and bone marrow function, in the absence of growth factors.
5. Fertility criteria:

   * Women of childbearing potential (WOCBP) and fertile males with WOCBP partners must use highly effective contraception
   * Women must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction
   * Men must agree not to donate sperm
   * A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a highly effective method of birth control.
6. Patient must be willing and able to adhere to the prohibitions and restrictions specified in the protocol. Due to the possibility of neurologic events, patient must agree to refrain from engaging in hazardous occupations or activities such as operating heavy or dangerous machinery during the first cycle of treatment.
7. Each patient must sign an informed consent form (ICF) indicating that he or she understands the purpose and procedures required for the study and is willing to participate in the study.

Exclusion Criteria:

1. Patient has any of the following medical situations:

   * Uncontrolled intercurrent illness including, but not limited to: poorly controlled hypertension; poorly controlled diabetes; ongoing active infection requiring antibiotics or acute infectious illness (including suspected viral infection); symptomatic congestive heart failure; unstable angina pectoris; cardiac arrhythmia considered to increase risk for the patient by the Investigator; psychiatric illness that would limit compliance with study requirement
   * Medical illness requiring systemic glucocorticoid use > 10mg/day prednisone equivalent.
   * Patients with any CNS disorder, such as CNS malignancy/metastasis, stroke, transient ischemic attack, or seizure disorder
   * Personal or familial history of hemophagocytic lymphohistiocytosis or macrophage activation syndrome
   * An autoimmune disease with a history of flares requiring immunosuppressant medications within the past 6 months
   * Prior allogeneic organ or bone marrow transplant (BMT).
   * Social situation that would limit compliance with study requirements
   * Major surgery (eg, requiring general anesthesia) within 4 weeks before the planned first dose of study drug, or not fully recovered from prior surgery, or has surgery planned during the time the patient is expected to participate in the study or within 4 weeks after the last dose of study drug.
   * History of positive testing for hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-hepatitis C virus) or other clinically active liver disease, or positive testing at screening for HBsAg or anti- hepatitis C virus.
   * History of human immunodeficiency virus (HIV) antibody positive
2. Patient has had prior therapy meeting the following:

   * Anticancer immunotherapy within 3 weeks prior to the first dose of CI-8993
   * Prior T Cell Receptor-modified or chimeric antigen receptor T cell (CART) therapy
   * Other anticancer therapy, including chemotherapy, targeted therapy, or treatment with an investigational anticancer agent within 2 weeks prior to the first dose of CI-8993
   * Radiotherapy (excluding limited palliative radiation) within 2 weeks of start of CI-8993
   * Unresolved toxicities from previous anticancer therapies above Grade 1.
   * Immune-related AE with prior immunotherapy that was Grade 3 or higher.
   * Patient has known allergies, hypersensitivity, or intolerance to components of CI 8993
3. Patient receiving therapeutic anticoagulants
4. Fertility exclusions:

   * Patient is pregnant, breastfeeding, or planning to become pregnant while enrolled in this study or within 3 months after the last dose of study drug; WOCBP must have a negative pregnancy status confirmed by serum pregnancy test at screening and within 72 hours of first dose of study drug.
   * Patient is a man who plans to father a child while enrolled in this study or within 3 months after the last dose of study drug.
5. Vaccinated with a live vaccine within 28 days (with the exception of the annual inactivated influenza vaccine) prior to the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of CI-8993 | 2 years
  The highest dose at a schedule, at which the DLT rate during the first cycle of this study (28 days from the first full dose) is < 33% in at least 6 patients.
Determine the Recommended Phase 2 dose (RP2D) | 2 years
  The RP2D will be a dose considered to be appropriately safe for a target phase 2 population and exhibit PK and PD characteristics that are favorable and considered likely to support clinical efficacy of CI-8993. The RP2D will be defined by the Safety Review Committee (SRC) based on PK, PD, safety, efficacy results in this study, as well as practical limitations.

SECONDARY OUTCOMES:
To characterize the pharmacokinetic (PK) parameters of CI-8993 measured by Cmax | 6 months
  maximum serum concentration (Cmax)
To characterize the pharmacokinetic (PK) parameters of CI-8993 measured by Cmin | 6 months
  trough serum concentration (Cmin)
To characterize the pharmacokinetic (PK) parameters of CI-8993 measured by Tmax | 6 months
  Time to maximum serum concentration
To characterize the pharmacokinetic (PK) parameters of CI-8993 measured by Area under the concentration versus time curve (AUC) | 6 months
  area under the concentration-time curve
To characterize the pharmacokinetic (PK) parameters of CI-8993 measured by T 1/2 | 6 months
  Serum terminal elimination half-life (T 1/2)
To characterize the pharmacokinetic (PK) parameters of CI-8993 measured by volume of distribution at steady state | 6 months
  volume of distribution at steady state (Vdss)
To characterize the pharmacokinetic (PK) parameters of CI-8993 measured by clearance | 6 months
  Clearance (CL)
To assess anti-drug antibodies (ADA) of CI-8993 | 6 months
  Evaluate antibodies to CI-8993 in serum
To assess objective response rate (ORR) | 2 years
  Assess with Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
To assess duration of response (DOR) | 2 years
  Assess with Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1 )
To evaluate safety of concomitant drugs that are cytochrome P450 (CYP) enzyme substrates with narrow therapeutic index and drug-drug interaction potential | 2 years
  An analysis of AEs considered related to concomitant drugs that are CYP enzyme substrates with narrow therapeutic index and drug-drug interaction potential

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Sarah Cannon Research Institute/Tennessee Oncology, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zong L, Mo S, Sun Z, Lu Z, Yu S, Chen J, Xiang Y. Analysis of the immune checkpoint V-domain Ig-containing suppressor of T-cell activation (VISTA) in endometrial cancer. Mod Pathol. 2022 Feb;35(2):266-273. doi: 10.1038/s41379-021-00901-y. Epub 2021 Sep 7. PMID 34493823